CLINICAL TRIAL: NCT00527397
Title: An Open-Label, Uncontrolled Long-Term Safety Study Of CP-464,005 (Inhaled Insulin) In Japanese Patients With Type 1 Or Type 2 Diabetes
Brief Title: Long-Term Safety Study Of Inhaled Insulin (CP-464,005, Inhaler) In Japanese Patients With Type1 or Type2 Diabetes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2171105
Record Dates: First submitted 2007-09-07; First posted 2007-09-10 (Estimated); Results first posted 2009-10-05 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-07

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Exubera

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- B (Experimental): Type 2 Diabetes Mellitus (DM) who has not yet treated by Insulin
  Interventions: Drug: CP-464,005
- C (Experimental): Type 2 DM who has already treated by Insulin
  Interventions: Drug: CP-464,005
- A (Experimental): Type 1 DM
  Interventions: Drug: CP-464,005

INTERVENTIONS:
Drug: CP-464,005 — Taken for 1 year (52 weeks) immediately before each meal (breakfast, lunch, and supper). Dose: adjusted based on the results of self-monitoring of blood glucose before each meal.
  Other Names: Exubera
  Arms: C
Drug: CP-464,005 — Taken for 1 year (52 weeks) immediately before each meal (breakfast, lunch, and supper). Dose: adjusted based on the results of self-monitoring of blood glucose before each meal.
  Other Names: Exubera
  Arms: A
Drug: CP-464,005 — Taken for 1 year (52 weeks) immediately before each meal (breakfast, lunch, and supper). Dose:adjusted based on the results of self-monitoring of blood glucose before each meal.
  Other Names: Exubera
  Arms: B

SUMMARY:
Assess the safety and toleration of CP-464,005 and Inhaler following 1-year (52 week) administration to Type 1 and Type 2 diabetes patients (non-smokers)

DETAILED DESCRIPTION:
Pfizer announced in October 2007 that it would stop marketing CP-464,005. At that time recruitment for study, A2171105 was placed on hold. Nektar, the company from which Pfizer licensed CP-464,005, announced on April 9, 2008 that it had stopped its search for a new marketing partner. As a result, study A2171105 was terminated on April 10, 2008. Neither safety nor efficacy reasons were the cause of the study termination.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed with Type 1 or Type 2 diabetes for at least 1 year, based on the diagnostic criteria for diabetes.

Exclusion Criteria:

* Patients who have smoked during the 6 months prior to screening (smoking shall be prohibited during the term of this study, as well)
* Patients exhibiting pulmonary function test (spirometry) abnormalities (FVC or FEV1 < 70% of predicted) ) at Week -4.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- Japan (10):
  - Pfizer Investigational Site, Nagoya, Aichi-ken
  - Pfizer Investigational Site, Yokohama, Kanagawa
  - Pfizer Investigational Site, Kyoto, Kyoto
  - Pfizer Investigational Site, Tenri-shi, Nara
  - Pfizer Investigational Site, Takatsuki-shi, Oosaka
  - Pfizer Investigational Site, Osaka, Osaka
  - Pfizer Investigational Site, Bunkyo-ku, Tokyo
  - Pfizer Investigational Site, Meguro-ku, Tokyo
  - Pfizer Investigational Site, Toyama, Toyama
  - Pfizer Investigational Site, Tokyo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2171105&StudyName=Long-Term%20Safety%20Study%20Of%20Inhaled%20Insulin%20%28CP-464%2C005%2C%20CP-464%2C005/Inhaler%29%20In%20Japanese%20Patients%20With%20Type1%20or%20Type2%20Diabetes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 centers in Japan.
Pre-assignment Details: As a result of Pfizer's decision (18 Oct 2007) to return the worldwide rights for CP-464,005 (insulin human [rDNA origin] Inhalation Powder) to Nektar, from which Pfizer licensed inhaled insulin technology, it was decided to terminate this study before it had recruited targeted number of subjects.
Groups:
- All Subjects With Type 1 or Type 2 Diabetes Mellitus: All subjects with type 1 or type 2 diabetes mellitus treated with inhaled insulin in this study. This study was open-label, uncontrolled study and at all times in the trial, each subject had an individualized recommended insulin dose for each of the dosing times.
Period: Overall Study
Arm/Group | All Subjects With Type 1 or Type 2 Diabetes Mellitus
Started | 24
Completed | 0
Not Completed | 24
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 6
Not completed — Study terminated by sponsor | 13

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects With Type 1 or Type 2 Diabetes Mellitus
Number analyzed (Participants) | 24
Age Continuous [Mean (Standard Deviation); unit: years] | 55.2 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 11

OUTCOME MEASURES:

1. Secondary Outcome: Daily Inhaled Insulin Dose
Description: The mean of daily inhaled insulin dose. The dose of inhaled insulin was adjusted based on the results of self-monitoring of blood glucose before each meal.The end of treatment values were calculated each subject's last observed value up to 26 weeks.
Time Frame: Up to 26 weeks
Population: Includes all subjects who received at least one dose of study drug. Number of subjects with evaluable data presented as n=type 1 Diabetes Mellitus, Type 2 Diabetes Mellitus Using Insulin, Type 2 Diabetes Mellitus Not Using Insulin, respectively.
Measure: Mean (Standard Deviation); unit: milligram
Groups:
- Type 1 Diabetes Mellitus: subjects with type 1 diabetes mellitus
- Type 2 Diabetes Mellitus Using Insulin: subjects with type 2 diabetes mellitus who had already treated by Insulin
- Type 2 Diabetes Mellitus Not Using Insulin: subjects with type 2 diabetes mellitus who had not yet treated by Insulin
Arm/Group | Type 1 Diabetes Mellitus | Type 2 Diabetes Mellitus Using Insulin | Type 2 Diabetes Mellitus Not Using Insulin
Number analyzed (Participants) | 6 | 12 | 6
milligram
  Day 1 (n=6, 12, 6) | 8.8 (3.4) | 7.2 (2.5) | 5.5 (2.3)
  Day 2 (n=6, 12, 6) | 9.7 (4.0) | 7.6 (3.5) | 5.5 (2.3)
  Day 3 (n=6, 12, 6) | 9.8 (4.6) | 7.8 (3.8) | 5.8 (2.5)
  Day 4 (n=6, 12, 6) | 10.0 (4.1) | 7.8 (3.8) | 5.5 (2.3)
  Day 5 (n=6, 12, 6) | 7.7 (3.7) | 7.8 (3.8) | 5.5 (2.6)
  Week 1 (n=6, 12, 6) | 9.8 (4.3) | 8.5 (5.0) | 5.8 (2.5)
  Week 2 (n=6, 11, 6) | 9.3 (3.9) | 8.9 (5.6) | 5.5 (2.9)
  Week 4 (n=5, 11, 6) | 8.4 (5.0) | 8.4 (5.1) | 5.2 (2.6)
  Week 6 (n=5, 9, 6) | 8.8 (4.3) | 8.1 (5.6) | 5.8 (2.9)
  Week 8 (n=5, 8, 6) | 8.0 (4.4) | 9.0 (6.6) | 5.7 (2.7)
  Week 12 (n=4, 7, 5) | 5.5 (1.7) | 9.9 (6.6) | 5.4 (3.0)
  Week 16 (n=3, 6, 3) | 6.0 (2.6) | 11.5 (7.7) | 5.0 (2.0)
  Week 20 (n=3, 5, 3) | 5.0 (2.0) | 12.4 (8.2) | 6.3 (1.5)
  Week 26 (n=3, 5, 3) | 6.0 (2.6) | 12.4 (8.2) | 6.3 (1.5)
  End of treatment (n=6, 12, 6) | 7.7 (4.0) | 9.1 (6.7) | 6.8 (2.6)

2. Secondary Outcome: The Values of Hemoglobin A1c:Change From Baseline
Description: Hemoglobin A1c levels obtained each observation point minus that at baseline. The end of treatment values were calculated each subject's last observed value up to 26 weeks.
Time Frame: Baseline, Week 6, Week 12, Week 26, End of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Type 1 Diabetes Mellitus | Type 2 Diabetes Mellitus Using Insulin | Type 2 Diabetes Mellitus Not Using Insulin
Number analyzed (Participants) | 6 | 12 | 6
percent
  Week 6 (n=5, 10, 6) | -0.42 (0.53) | -0.39 (0.55) | -0.72 (1.09)
  Week 12 (n=4, 6, 3) | -0.35 (0.76) | -0.48 (0.72) | -0.93 (0.38)
  End of treatment (n=6, 12, 6) | -0.22 (0.90) | 0.01 (0.78) | -0.48 (1.20)

3. Secondary Outcome: The Value of Fasting Plasma Glucose:Change From Baseline
Description: Fasting plasma glucose levels obtained at each observation point minus that at baseline. The end of treatment values were calculated each subject's last observed value up to 26 weeks.
Time Frame: Baseline, Week 6, Week 12, Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligram/millilitre
Arm/Group | Type 1 Diabetes Mellitus | Type 2 Diabetes Mellitus Using Insulin | Type 2 Diabetes Mellitus Not Using Insulin
Number analyzed (Participants) | 6 | 12 | 6
milligram/millilitre
  Week 6 (n=4, 10, 6) | 50.3 (31.3) | -1.6 (96.4) | -3.0 (39.0)
  Week 12 (n=3, 6, 3) | 27.7 (27.1) | 11.3 (47.9) | -5.0 (16.5)
  End of treatment (n=4, 12, 6) | 87.3 (83.0) | 18.3 (76.9) | -8.8 (47.9)

4. Secondary Outcome: The Incidence of Hypoglycaemia at the Cumulative Doses of Inhaled Insulin
Description: Number of hypoglycemic events per subject-month. Subject-month=(number of days from the first day of study treatment to the last day of active treatment + 1 day lag)/30.44
Time Frame: 0 month to 12 months
Population: as for outcome 1
Measure: Number; unit: events / subject-month
Arm/Group | Type 1 Diabetes Mellitus | Type 2 Diabetes Mellitus Using Insulin | Type 2 Diabetes Mellitus Not Using Insulin
Number analyzed (Participants) | 6 | 12 | 6
events / subject-month
  0 to 3 months (n=6, 12, 6) | 3.5 | 3.2 | 0.1
  >3 to 6 months (n=3, 6, 4) | 0.1 | 0.2 | 0.3
  overall (n=6, 12, 6) | 1.9 | 1.9 | 0.2

5. Secondary Outcome: The Values of Forced Expiratory Volume at 1 Second:Change From Baseline
Description: Pulmonary function test(forced expiratory volume at 1 second) obtained at each observation point minus that at baseline. The end of treatment values were calculated each subject's last observed value up to 26 weeks.
Time Frame: Beseline, Week 1, Week 2, Week 6, Week 12, Week 26
Population: Included all subjects who had a baseline forced expiratory volume at 1 second value, had at least one-post baseline forced expiratory volume at 1 second values, and received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: liter
Groups:
- All Subjects: subjects treated with inhaled insulin
Arm/Group | All Subjects
Number analyzed (Participants) | 24
liter
  Week 1 (n=23) | -0.055 (0.162)
  Week 2 (n=22) | -0.070 (0.184)
  Week 6 (n=21) | -0.065 (0.126)
  Week 12 (n=13) | 0.012 (0.137)
  Week 26 (n=4) | -0.030 (0.086)
  End of treatment (n=24) | -0.034 (0.147)

6. Secondary Outcome: The Values of Forced Vital Capacity:Change From Baseline
Description: pulmonary function test(forced vital capacity) obtained at each observation point minus that at baseline. The end of treatment values were calculated each subject's last observed value up to 26 weeks.
Time Frame: Baseline, Week 1, Week 2, Week 6, Week 12, Week 26, End of treatment
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | All Subjects
Number analyzed (Participants) | 24
liter
  Week 1 (n=23) | -0.053 (0.208)
  Week 2 (n=22) | 0.000 (0.135)
  Week 6 (n=21) | -0.003 (0.176)
  Week 12 (n=13) | 0.065 (0.204)
  Week 26 (n=4) | -0.105 (0.074)
  End of treatment (n=24) | -0.001 (0.169)

7. Secondary Outcome: The Values of Forced Expiratory Volume at 1 Second/Forced Vital Capacity:Change From Baseline
Description: Pulmonary function test(forced expiratory volume at 1 second/forced vital capacity) obtained at each observation point minus that at baseline. The end of treatment values were calculated each subject's last observed value up to 26 weeks.
Time Frame: Baseline, Week 1, Week 2, Week 6, Week 12, Week26, End of treatment
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: liter/liter
Arm/Group | All Subjects
Number analyzed (Participants) | 24
liter/liter
  Week 1 (n=23) | -0.003 (0.033)
  Week 2 (n=22) | -0.023 (0.038)
  Week 6 (n=21) | -0.022 (0.034)
  Week 12 (n=13) | -0.012 (0.029)
  Week 26 (n=4) | 0.013 (0.013)
  End of treatment (n=24) | -0.012 (0.043)

8. Secondary Outcome: Insulin Antibody Levels : Change From Baseline
Description: Insulin antibody levels obtained at each observation point minus that at baseline. The end of treatment values were calculated each subject's last observed value up to 26 weeks.
Time Frame: Baseline, Week 6, Week 12, End of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microunit/milliliter
Arm/Group | Type 1 Diabetes Mellitus | Type 2 Diabetes Mellitus Using Insulin | Type 2 Diabetes Mellitus Not Using Insulin
Number analyzed (Participants) | 6 | 12 | 6
microunit/milliliter
  Week 6 (n=5, 10, 6) | 1.68 (5.71) | 3630.63 (11026.91) | -0.42 (5.40)
  Week 12 (n=4, 6, 3) | 9.78 (7.02) | 131.73 (154.02) | 11.00 (14.29)
  End of treatment (n=6, 12, 6) | 10.52 (11.49) | 3220.95 (10025.38) | 11.42 (9.04)

9. Primary Outcome: Self-Monitoring Blood Glucose Levels: Change From Baseline
Description: Self-monitoring blood glucose levels obtained at each observation point minus that at baseline.
Time Frame: One year
Population: This endopoint was not analyzed because of small numbers of subjects due to early termination
Measure: Mean (Standard Deviation); unit: milligram/millilitre
Arm/Group | Type 1 Diabetes Mellitus | Type 2 Diabetes Mellitus Using Insulin | Type 2 Diabetes Mellitus Not Using Insulin
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | All Subjects With Type 1 or Type 2 Diabetes Mellitus
Serious Adverse Events (participants affected / at risk) | 3
Other Adverse Events (participants affected / at risk) | 23
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | All Subjects With Type 1 or Type 2 Diabetes Mellitus
Tendon rupture (Injury, poisoning and procedural complications) | 1/24
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1/24
Hyperglycaemia (Metabolism and nutrition disorders) | 1/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | All Subjects With Type 1 or Type 2 Diabetes Mellitus
Diarrhoea (Gastrointestinal disorders) | 2/24
Hunger (General disorders) | 2/24
Nasopharyngitis (Infections and infestations) | 7/24
Tinea pedis (Infections and infestations) | 2/24
Device malfunction (Injury, poisoning and procedural complications) | 4/24
Urine ketone body present (Investigations) | 2/24
Hypoglycaemia (Metabolism and nutrition disorders) | 16/24
Dizziness (Nervous system disorders) | 2/24
Cough (Respiratory, thoracic and mediastinal disorders) | 4/24
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2/24

LIMITATIONS AND CAVEATS:
As a result of Pfizer's decision (18 Oct 2007) to return the worldwide rights for CP-464,005 (insulin human [rDNA origin]) Inhalation Powder) to Nektar, from which Pfizer licensed inhaled insulin technology, it was decided to terminate this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.